CLINICAL TRIAL: NCT02887612
Title: A Prospective Study of Blood Circulating Tumor DNA for the Prediction of Postoperative Relapse in Early and Intermediate-Stage Gastric Cancer
Brief Title: ctDNA for Prediction of Relapse in Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, MD.,PhD., Sun Yat-sen University
Other Study IDs: ctDNA001
Record Dates: First submitted 2016-05-14; First posted 2016-09-02 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: ctDNA test

SUMMARY:
Gastric cancer is one of the common malignant tumors in China, with relatively high incident rate and mortality among the population. Surgery is the conventional treatment option for early and intermediate-stage stage gastric cancer, but postoperative relapse is the major issue. Circulating tumor DNA (ctDNA) is tumor-derived fragmented DNA with an average size of 166 bp, mixed with cell free DNA (cfDNA) of other sources in blood circulation.ctDNA is reflecting the most up-to-date status of tumor genome. Hence, it is considered as a new biomarker for tumor, which can be qualitative, quantitative and used for disease monitoring. The present clinical trial aims to elucidate the correlation between the serum ctDNA status and the prognosis of patients with early and intermediate-stage gastric cancer upon surgical treatment, and explore the possibility of clinical utility of serum ctDNA as a clinical index to predict postoperative relapse.

DETAILED DESCRIPTION:
Gastric cancer is one of the common malignant tumors in China, withrelatively high incident rate and mortality among the population. 95% of the gastric cancer is adenocarcinoma. 70% of the patients at the early stage show no obvious symptom, and only small number of them has nausea, vomiting, or symptoms that are similar to the of peptic ulcer disease.

Surgery is the conventional treatment option for early and middle stage gastric cancer, but postoperative relapse is the major issue. Currently, the only proven effective chemotherapies for gastric cancer are the taxane and platinum-based combination therapies. Also due to its molecular heterogeneity, the prognosis of gastric caner is highly varied among the patients. Therefore,there are not many effective targeting therapies available for the treatment of gastric cancer; and currently, trastuzumab and apatinib are the only two targeting drugs that have been clinically approved by CFDA.

Circulating tumor DNA (ctDNA) is tumor-derived fragmented DNA with an average size of 166 bp, mixed with cell free DNA (cfDNA) of other sources in blood circulation (2, 3). Although the mechanisms of its release have not been fully addressed, most reports considered apoptosis and/or necrosis of tumor cells as its main sources, which makes it a genomic reservoir of different tumor clones (4). Also, as its half-life is up to hours, ctDNA is reflecting the most up-to-date status of tumor genome(5). Hence, it is considered as a new biomarker for tumor, which can be qualitative, quantitative and used for disease monitoring.

By monitoring the serum ctDNA mutational profile using Next Generation Sequencing (NGS), the present clinical trial aims to elucidate the correlation between the serum ctDNA status and the prognosis of patients with early and intermediate-stage gastric cancer upon surgical treatment, and explore the possibility of clinical utility of serum ctDNA as a clinical index to predict postoperative relapse. Moreover, by comparing the molecular profiles of patients with different prognosis, we may also screen out the molecular markers related to the prognosis of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age at first visit.
2. Patients must have histologically confirmed early or intermediate-stage gastric cancer.
3. Patients need to have surgical treatment.
4. Patients must be able to provide sufficient fresh tissue/biopsies or minimum 5-10 FFPE sections for NGS analysis.
5. Patients must be able to follow the study visit schedule and willing to provide peripheral blood samples at the indicated time point.
6. Written informed consent must be obtained from patient or patient's legal representative and ability for patient to comply with the requirements of the study.

Exclusion Criteria:

1. Patients who cannot provide peripheral blood samples prior to the surgical treatment will be excluded.
2. Patients with severe infection will be excluded.
3. Patients with other serious disease besides early or intermediate-stage gastric cancer will be excluded.
4. Pregnant women will be excluded.
5. Patients who are alcoholic or drug abusers will be excluded.
6. Patients with a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective clinical study collaborated with Geneseeq Technology Inc.200 of patients are planned. Total duration of the study is expected to be 2 years. The fresh tumor tissues/biopsies of each patient will be collected during the surgical treatment. The peripheral blood samples of each patient will be collected at the following time points: 1) prior to the surgical treatment; 2) 1 week after the surgical treatment; 3)every three months until disease progression or the end of the study. The collected fresh tumor tissues/biopsies or formalin fixed paraffin embedded (FFPE) blocks/sections, and peripheral blood samples will be further subjected for NGS analysis and NGS-based ctDNA mutation profiling, respectively.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value | through study completion, an average of 2 years
  the proportions of patients with positive serum ctDNA (in any follow-up) that have postoperative relapse

SECONDARY OUTCOMES:
prognostic molecular markers | through study completion, an average of 2 years
  to screen out the molecular markers related to the prognosis of gastric cancer by comparing the molecular profiles of patients with different prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Medical Oncology,Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jahr S, Hentze H, Englisch S, Hardt D, Fackelmayer FO, Hesch RD, Knippers R. DNA fragments in the blood plasma of cancer patients: quantitations and evidence for their origin from apoptotic and necrotic cells. Cancer Res. 2001 Feb 15;61(4):1659-65. PMID 11245480
- [Background] Jiang P, Chan CW, Chan KC, Cheng SH, Wong J, Wong VW, Wong GL, Chan SL, Mok TS, Chan HL, Lai PB, Chiu RW, Lo YM. Lengthening and shortening of plasma DNA in hepatocellular carcinoma patients. Proc Natl Acad Sci U S A. 2015 Mar 17;112(11):E1317-25. doi: 10.1073/pnas.1500076112. Epub 2015 Feb 2. PMID 25646427
- [Background] Stroun M, Lyautey J, Lederrey C, Olson-Sand A, Anker P. About the possible origin and mechanism of circulating DNA apoptosis and active DNA release. Clin Chim Acta. 2001 Nov;313(1-2):139-42. doi: 10.1016/s0009-8981(01)00665-9. PMID 11694251
- [Background] Yu SC, Lee SW, Jiang P, Leung TY, Chan KC, Chiu RW, Lo YM. High-resolution profiling of fetal DNA clearance from maternal plasma by massively parallel sequencing. Clin Chem. 2013 Aug;59(8):1228-37. doi: 10.1373/clinchem.2013.203679. Epub 2013 Apr 19. PMID 23603797
- [Derived] Yuan SQ, Nie RC, Huang YS, Chen YB, Wang SY, Sun XW, Li YF, Liu ZK, Chen YX, Yao YC, Xu Y, Qiu HB, Liang Y, Wang W, Liu ZX, Zhao Q, Xu RH, Zhou ZW, Wang F. Residual circulating tumor DNA after adjuvant chemotherapy effectively predicts recurrence of stage II-III gastric cancer. Cancer Commun (Lond). 2023 Dec;43(12):1312-1325. doi: 10.1002/cac2.12494. Epub 2023 Oct 14. PMID 37837629